CLINICAL TRIAL: NCT03940508
Title: Engaging Black Youth in Depression and Suicide Prevention Treatment Within Urban Schools: A Preliminary Study
Brief Title: Engaging Black Youth in Depression and Suicide Prevention Treatment Within Urban Schools
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: New York University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH); Columbia University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1R34MH119290-01 (NIH); 1R34MH119290-01 (NIH)
Record Dates: First submitted 2019-04-29; First posted 2019-05-07 (Actual); Results first posted 2025-09-15 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2023-09

CONDITIONS: Depression; Suicidal Ideation
Keywords: depression; treatment engagement; adolescents; Black youth; Intervention
MeSH Terms: conditions — Depression; Suicidal Ideation | interventions — Interpersonal Psychotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MCI + IPT-A (Experimental): Participants will receive the Making Connections Intervention (MCI) in addition to IPT-A for depression.
  Interventions: Behavioral: Making Connections Intervention; Behavioral: IPT-A
- IPT-A Only (Active Comparator): Participants will receive IPT-A for depression.
  Interventions: Behavioral: IPT-A

INTERVENTIONS:
Behavioral: Making Connections Intervention — The MCI is a one to two session intervention that addresses barriers to mental health treatment and helps adolescents build skills to get the most out of their treatment experience. It is designed to be delivered by a trained clinician in conjunction with an evidence-based treatment.
  Arms: MCI + IPT-A
Behavioral: IPT-A — IPT-A is a time-limited, manualized treatment for depression focused on maladaptive communication patterns and interpersonal interactions.
  Other Names: Interpersonal Psychotherapy for Depressed Adolescents

SUMMARY:
Completing evidence-based treatments for depression has been shown to be particularly problematic for Black adolescents. If Black adolescents' depression treatment needs are to be met, the engagement challenges and the factors that lessen the success of treatment in the "real world" must be addressed. The investigators will examine the effectiveness of the Making Connections Intervention (MCI) and investigate key mediators of both engagement and response to treatment for depression. The MCI is a 1-2 session, evidence-based intervention designed to improve engagement, perceived relevance, and treatment satisfaction among depressed, Black adolescents. The study also uses tailored outreach strategies for adolescents and parents by including innovative digital content such as a web page/app along with other digital products.

This study will address an important public health issue: How best to connect Black adolescents with depression to treatment in clinically meaningful ways, and how best to deliver evidence-based treatment to them through school-based services.

DETAILED DESCRIPTION:
Completing evidence-based treatments for depression has been shown to be particularly problematic for Black adolescents. Their rates of participation in treatments for depression are lower due to negative perceptions of services and providers, and their reluctance to acknowledge the presence of symptoms.

If Black adolescents' depression treatment needs are to be met, the engagement challenges and the factors that lessen the success of treatment in the "real world" must be addressed. This research examines the effectiveness of the Making Connections Intervention (MCI) and investigates key mediators of both engagement and response to treatment for depression. The MCI is a 1-2 session, evidence-based intervention designed to improve engagement, perceived relevance, and treatment satisfaction among depressed, Black adolescents. The study also uses tailored outreach strategies for adolescents and parents by including innovative digital content such as a web page/app along with other digital products.

The investigators previously performed a small pilot study that used the MCI as an add-on to the IPT-A, an evidence-based intervention for depression delivered in schools typically over 12 sessions. The results suggested that MCI has a positive impact on many aspects of change associated with treatment engagement and clinical outcomes.

This study will be a randomized controlled trial. It will examine the effectiveness of the MCI in a multi-school trial involving adolescents in grades 6-12 who attend New York City (NYC) Department of Education (DOE) Public Schools. The investigators will randomly assign 60 Black students with depression symptoms to two conditions: MCI+IPT-A vs. IPT-A-alone. The investigators will also do qualitative research, like interviews, before the digital content is created. This will enhance the relevance of the MCI. The main outcomes are adolescent-and caregiver-level engagement and adolescent depression. Suicidal ideation is a secondary outcome. This study will also test related factors, like adolescent helping-seeking behavior and parental knowledge of mental health services, that can account for treatment outcomes and that will allow the MCI to be strengthened in future roll-outs of the intervention in school settings.

ELIGIBILITY:
Inclusion Criteria:

1. Must identify as Black and/or African American
2. Must be enrolled in grades 6-12 (except 12th graders in their last semester)
3. Must be able to speak English
4. Must have received caregiver consent and have assented to participate
5. Must meet depression and global functioning levels indicated by a CES-D score ≥16, a Hamilton Rating Scale of Depression (HRSD) Score ≥ 10, and a Global Assessment Scale for Children (C-GAS) score ≤ 65 at baseline
6. Students who are currently on a stable dose of anti-depressant medication, but still meet inclusion criteria, can be enrolled in the study.

Exclusion Criteria:

1. Actively suicidal with intent or plan
2. Intellectually disabled
3. Have a life threatening medical illness
4. Have a current primary substance abuse diagnosis in the moderate to severe range, schizophrenia, bipolar disorder, any evidence of psychosis, a primary diagnosis of anorexia
5. Currently in active treatment for depression (excluding medication) at baseline assessment

Ages: 12 Years to 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 29 (Actual)
Dates: Start 2020-01-31 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael A Lindsey, PhD, Principal Investigator — NYU Silver School of Social Work
Locations (2):
- United States (2):
  - Columbia University, New York, New York
  - McSilver Institute for Poverty Policy and Research, New York, New York

IPD SHARING:
Plan to Share IPD: Yes
Submit data in compliance with NIMH Data Archive data submission agreement.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: By the end of data collection, December 2023.
Access Criteria: In accordance with the NIMH Data Archive requirements.

REFERENCES:
- [Background] Gunlicks-Stoessel M, Mufson L, Jekal A, Turner JB. The impact of perceived interpersonal functioning on treatment for adolescent depression: IPT-A versus treatment as usual in school-based health clinics. J Consult Clin Psychol. 2010 Apr;78(2):260-7. doi: 10.1037/a0018935. PMID 20350036
- [Background] Mufson L, Moreau D, Weissman MM, Wickramaratne P, Martin J, Samoilov A. Modification of interpersonal psychotherapy with depressed adolescents (IPT-A): phase I and II studies. J Am Acad Child Adolesc Psychiatry. 1994 Jun;33(5):695-705. doi: 10.1097/00004583-199406000-00011. PMID 8056733
- [Background] Mufson LH, Dorta KP, Olfson M, Weissman MM, Hoagwood K. Effectiveness research: transporting interpersonal psychotherapy for depressed adolescents (IPT-A) from the lab to school-based health clinics. Clin Child Fam Psychol Rev. 2004 Dec;7(4):251-61. doi: 10.1007/s10567-004-6089-6. PMID 15648279
- [Background] Lindsey MA, Chambers K, Pohle C, Beall P, Lucksted A. Understanding the Behavioral Determinants of Mental Health Service Use by Urban, Under-Resourced Black Youth: Adolescent and Caregiver Perspectives. J Child Fam Stud. 2013 Jan 1;22(1):107-121. doi: 10.1007/s10826-012-9668-z. Epub 2012 Oct 16. PMID 23355768
- [Background] Lindsey MA, Joe S, Nebbitt V. Family Matters: The Role of Mental Health Stigma and Social Support on Depressive Symptoms and Subsequent Help Seeking Among African American Boys. J Black Psychol. 2010 Nov 1;36(4):458-482. doi: 10.1177/0095798409355796. PMID 20953336
- [Background] Breland-Noble AM, Bell CC, Burriss A; AAKOMA Project Adult Advisory Board. "Mama just won't accept this": adult perspectives on engaging depressed African American teens in clinical research and treatment. J Clin Psychol Med Settings. 2011 Sep;18(3):225-34. doi: 10.1007/s10880-011-9235-6. PMID 21512751
- [Background] Lindsey MA, Korr WS, Broitman M, Bone L, Green A, Leaf PJ. Help-seeking behaviors and depression among African American adolescent boys. Soc Work. 2006 Jan;51(1):49-58. doi: 10.1093/sw/51.1.49. PMID 16512510
- [Background] Lindsey MA, Brown DR, Cunningham M. Boys do(n't) cry: Addressing the unmet mental health needs of African American boys. Am J Orthopsychiatry. 2017;87(4):377-383. doi: 10.1037/ort0000198. PMID 28691838
- [Background] Ellis ML, Lindsey MA, Barker ED, Boxmeyer CL, Lochman JE. Predictors of engagement in a school-based family preventive intervention for youth experiencing behavioral difficulties. Prev Sci. 2013 Oct;14(5):457-67. doi: 10.1007/s11121-012-0319-9. PMID 23420474
- [Derived] Lindsey MA, Mufson L, Velez-Grau C, Grogan T, Wilson DM, Reliford AO, Gunlicks-Stoessel M, Jaccard J. Engaging Black youth in depression and suicide prevention treatment within urban schools: study protocol for a randomized controlled pilot. Trials. 2024 Feb 9;25(1):112. doi: 10.1186/s13063-024-07947-8. PMID 38336803
- See also: Lu W, Lindsey M, Irsheid S, Nebbitt V. Psychometric properties of the center for epidemiological studies-depression Scale (CES-D) among Black adolescents. Journal of the Society for Social Work and Research. 2017. — https://www.journals.uchicago.edu/doi/full/10.1086/694791#

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | MCI + IPT-A | IPT-A Only
Started | 19 | 10
Completed | 9 | 2
Not Completed | 10 | 8

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | MCI + IPT-A | IPT-A Only | Total
Number analyzed (Participants) | 19 | 10 | 29
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 17 | 10 | 27
  Between 18 and 65 years | 2 | 0 | 2
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: Months] | 194.68 (17.29) | 193.80 (11.51) | 194.37 (15.32)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 10 | 23
  Male | 6 | 0 | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 19 | 10 | 29
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 19 | 10 | 29

OUTCOME MEASURES:

1. Primary Outcome: Center for Epidemiological Studies-Depression Scale
Description: A 20-item self-report scale designed to measure depressive symptomatology in the general population. Scores range from 0 to 60, with higher scores indicating greater depression symptoms. 16 is a common clinical cutoff.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | MCI + IPT-A | IPT-A Only
Number analyzed (Participants) | 19 | 10
units on a scale | 36.84 (11.85) | 40.90 (11.60)

2. Primary Outcome: Hamilton Rating Scale for Depression
Description: Determines a patient's level of depression before, during, and after treatment. Scores range from 0 to 52, with higher scores indicating greater severity of depression. Scores of 0-7 indicate no depression.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | MCI + IPT-A | IPT-A Only
Number analyzed (Participants) | 19 | 10
units on a scale | 14.47 (8.66) | 16.60 (7.33)

3. Primary Outcome: Demographic Form
Description: To measure participants' demographic characteristics
Time Frame: Baseline
Measure: Number; unit: participants
Arm/Group | MCI + IPT-A | IPT-A Only
Number analyzed (Participants) | 19 | 10
participants
  Born in NYC-Yes | 17 | 9
  Born in NYC-No | 2 | 1
  Sex-Female | 13 | 10
  Sex-Male | 6 | 0
  Disability-Yes | 0 | 1
  Special Education-Yes | 0 | 1
  Ever treatment for emotional or behavioral difficulties?-Yes | 3 | 1

4. Primary Outcome: Columbia-Suicide Severity Rating Scale
Description: To assess the severity and lethality of suicidal behaviors and ideations, and can be used to monitor treatment outcomes and establish suicide risk in a variety of research and clinical settings. "Yes" and "No" categories are used to determine suicide risk, with binary coding where No=0 and Yes=1 for items 1-5. The higher number indicating more intense ideation. Total scores of items 1-5 were analyzed, with the lowest score =0 and the highest score=5.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | MCI + IPT-A | IPT-A Only
Number analyzed (Participants) | 19 | 10
units on a scale | 0.94 (1.68) | 1.1 (2.13)

5. Primary Outcome: Barriers for Adolescents Seeking Health
Description: Self-report questionnaire that targets barriers to seeking professional psychological help. Scores range from 37 to 111, with higher scores indicating greater barriers to help seeking behaviors.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | MCI + IPT-A | IPT-A Only
Number analyzed (Participants) | 19 | 10
units on a scale | 62.52 (4.56) | 66.5 (5.42)

6. Primary Outcome: Child Help-Seeking Scale
Description: Self-report 28-item questionnaire designed to measure children's and adolescents' willingness to seek help for psychosocial problems from adults in the school setting. Scores for part one range from 16 to 64 and scores for part two rang from 7 to 28, with higher scores indicating less help- seeking.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | MCI + IPT-A | IPT-A Only
Number analyzed (Participants) | 19 | 10
units on a scale
  HSS Part 1 | 38.68 (3.62) | 39.6 (2.67)
  HSS Part 2 | 16.78 (5.22) | 16.44 (4.8)

7. Primary Outcome: Attitudes Toward Psychological Help Scale
Description: This scale assesses psychological factors, including stigma, perceived relevance of treatment, etc., that impact one's perceptions of and attitudes about using formal mental health treatment services. Scores range from 0-15, with higher scores indicating greater stigma.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | MCI + IPT-A | IPT-A Only
Number analyzed (Participants) | 19 | 10
units on a scale | 6.21 (3.04) | 6.8 (2.14)

8. Primary Outcome: Stages of Change
Description: 32-item instrument for assessing the readiness for changes in relation to general problems, or problems associated with participation in psychotherapy. The highest score among each sub-scale indicates which stage of change a person is in. Thus, sub-scale scores are reported. Sub-scale scores do not indicate a better or worse outcome; instead, higher scores indicate a readiness to take action to address mental health concerns on each sub-scale. Pre-contemplation scores range from 5-20, Contemplation scores range from 4-16, Action scores range from 5-20, and Maintenance scores range from 4-16.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | MCI + IPT-A | IPT-A Only
Number analyzed (Participants) | 19 | 10
units on a scale
  Pre-contemplation | 9.78 (1.87) | 9.8 (2.52)
  Contemplation | 13.05 (1.39) | 13.5 (1.43)
  Action | 15.26 (2.02) | 14.5 (3.27)
  Maintenance | 12.42 (2.34) | 12.4 (1.07)

9. Primary Outcome: Barriers to Treatment Participation Scale
Description: To test whether perceived barriers to treatment influence dropping out and other measures of participation in treatment. To assess a broad range of barriers evident over the course of treatment, including four thematic areas: stressors and obstacles that compete with treatment, treatment demands and issues, perceived relevance of treatment, and relationship with the therapist. Higher scores indicating greater barriers to treatment. Sub-scale scores range from 20 to 100 (Stressors), 10-50 (Demands), and 8-40 (Perceived Relevance of Treatment).
Time Frame: Baseline
Population: Caregiver measure
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | MCI + IPT-A | IPT-A Only
Number analyzed (Participants) | 15 | 7
units on a scale
  Total | 64.6 (25.85) | 54.14 (15.29)
  Subscale 1 (Stressors) | 35.06 (14.52) | 27.28 (7.06)
  Subscale 2 (Treatment Demands) | 16.46 (7.20) | 13.42 (5.59)
  Subscale 3 (Perceived Relevance of Treatment) | 13.06 (5.73) | 13.42 (4.27)

10. Primary Outcome: Understanding Mood Disorders Questionnaire
Description: Designed to measure family members' attributions about and knowledge of symptoms, course, and treatment of mood disorders. Scores range from 9 to 40, with higher scores indicating less understanding of how depression presents and functions.
Time Frame: Baseline
Population: Caregiver measure
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | MCI + IPT-A | IPT-A Only
Number analyzed (Participants) | 15 | 7
units on a scale | 18.73 (5.16) | 17 (3.65)

11. Primary Outcome: Therapy Survey
Description: To measure change in expectations about treatment at a children's psychiatric clinic about a week before their first therapy and counseling sessions. Scores range from 7 to 35, with higher scores indicating misconceptions about the role of therapy.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | MCI + IPT-A | IPT-A Only
Number analyzed (Participants) | 19 | 10
units on a scale | 14.8 (4.95) | 12.14 (3.8)

12. Primary Outcome: Suicidal Ideation Questionnaire-Junior
Description: A 15-item self-report measure developed specifically for identifying and assessing current suicidal ideation among young adolescents that requires approximately five to eight minutes to complete. Scores range from 0 to 90, with a typical clinical cutoff score of 31 indicating further evaluation due to increased risk of suicidal ideation.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | MCI + IPT-A | IPT-A Only
Number analyzed (Participants) | 19 | 10
units on a scale | 25.68 (17.01) | 29.3 (19.05)

13. Primary Outcome: Global Assessment Scale for Children
Description: To reflect the lowest level of functioning for a child or adolescent during a specified time period, or on a hypothetical continuum of health-illness. Higher scores indicate higher functioning, ranging from 1-100.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | MCI + IPT-A | IPT-A Only
Number analyzed (Participants) | 19 | 10
units on a scale | 57.84 (6.3) | 53.7 (7.42)

14. Primary Outcome: Interpersonal Needs
Description: A 15-item questionnaire to measure changes in students' social connectedness and social competence. Total scores ranging from 15-99 are reported with higher scores indicated less social connectedness.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | MCI + IPT-A | IPT-A Only
Number analyzed (Participants) | 19 | 10
units on a scale | 51.26 (13.55) | 61.5 (15.09)

15. Primary Outcome: Penn Helping Alliance Revised
Description: This questionnaire collects data from both the therapist and patient to measure the strength of the bond between therapist and patient, called the therapeutic alliance. Scores range from 6 to 36, with a higher score indicating greater therapeutic alliance.
Time Frame: Week 4
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | MCI + IPT-A | IPT-A Only
Number analyzed (Participants) | 8 | 5
units on a scale | 30.87 (3.76) | 29.2 (5.63)

ADVERSE EVENTS:
Time Frame: Baseline
Description: Any untoward medical occurrence associated in humans, whether or not considered treatment related.
Groups:
- MCI + IPT-A: Participants will receive the Making Connections Intervention (MCI) in addition to IPT-A for depression.
  Making Connections Intervention: The MCI is a one to two session intervention that addresses barriers to mental health treatment and helps adolescents build skills to get the most out of their treatment experience. It is designed to be delivered by a trained clinician in conjunction with an evidence-based treatment.
  IPT-A: IPT-A is a time-limited, manualized treatment for depression focused on maladaptive communication patterns and interpersonal interactions.
  No participants in our small sample experienced SAEs or AEs in either condition.
- IPT-A Only: Participants will receive IPT-A for depression.
  IPT-A: IPT-A is a time-limited, manualized treatment for depression focused on maladaptive communication patterns and interpersonal interactions.
  No participants in our small sample experienced SAEs or AEs in either condition.
Arm/Group | MCI + IPT-A | IPT-A Only
All-Cause Mortality (participants affected / at risk) | 0/19 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/10
Other Adverse Events (participants affected / at risk) | 0/19 | 0/10

LIMITATIONS AND CAVEATS:
Our recruitment was negatively impacted by COVID-19 and the closure of NYC Schools during the time of the study. While the study team pivoted to virtual recruitment and implementation, our inability to be onsite drastically reduced our ability to build rapport and recruit participants, yielding only 2 participants who completed IPT-A only and 9 who completed MCI+IPT-A. Baseline descriptives are reported only; the small sample size restricted our ability to compare groups on the outcome data.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2019-04-17): https://cdn.clinicaltrials.gov/large-docs/08/NCT03940508/Prot_000.pdf
  • Statistical Analysis Plan (2021-06-28): https://cdn.clinicaltrials.gov/large-docs/08/NCT03940508/SAP_001.pdf